CLINICAL TRIAL: NCT01440322
Title: AIR OPTIX® COLORS Registration Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CIBA VISION (Industry)
Responsible Party: Sponsor
Organization: Alcon Research (Industry)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: P-383-C-003 (C-11-032)
Record Dates: First submitted 2011-09-22; First posted 2011-09-26 (Estimated); Results first posted 2014-03-28 (Estimated); Last update posted 2014-05-08 (Estimated); Status verified 2014-04

CONDITIONS: Refractive Error
Keywords: Myopia; Contact lenses
MeSH Terms: conditions — Refractive Errors; Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AIR OPTIX® COLORS (Experimental): Lotrafilcon B contact lenses with color worn in both eyes on a daily wear, monthly replacement basis for 3 months
  Interventions: Device: Lotrafilcon B contact lens with color
- AIR OPTIX® AQUA (Active Comparator): Lotrafilcon B contact lenses worn in both eyes on a daily wear, monthly replacement basis for 3 months
  Interventions: Device: Lotrafilcon B contact lens

INTERVENTIONS:
Device: Lotrafilcon B contact lens with color — Silicone hydrogel contact lens with color
  Other Names: AIR OPTIX® COLORS
  Arms: AIR OPTIX® COLORS
Device: Lotrafilcon B contact lens — Silicone hydrogel contact lens
  Other Names: AIR OPTIX® AQUA
  Arms: AIR OPTIX® AQUA

SUMMARY:
The purpose of this study was to evaluate the subjective and objective performance and the physiological response to AIR OPTIX® COLORS soft contact lenses compared with AIR OPTIX® AQUA contact lenses in participants with normal eyes and prescription needs.

DETAILED DESCRIPTION:
This study consisted of 7 scheduled visits conducted over a 3-month period. Enrolled participants were randomized (2:1) to receive either AIR OPTIX® COLORS lenses in both eyes or AIR OPTIX® AQUA lenses in both eyes.

ELIGIBILITY:
Inclusion Criteria:

* Be of legal age of consent and sign Informed Consent document. If under legal age of consent, legally authorized representative must sign Informed Consent document and subject must sign Assent document.
* Normal eyes and not using any ocular medications.
* Willing to wear visitint or gray-colored spherical contact lenses in both eyes within available power ranges.
* Manifest cylinder less than or equal to 0.75 diopter.
* Best spectacle corrected visual acuity greater than or equal to 20/25.
* Have current prescription glasses.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Anterior segment infection, inflammation, or abnormality.
* Any active anterior segment ocular or systemic disease that would contraindicate contact lens wear.
* Use of ocular or systemic medications for which contact lens wear could be contraindicated as determined by the investigator.
* History of refractive surgery or irregular cornea.
* History of pathologically dry eye.
* Corneal vascularization greater than 1 millimeter of penetration.
* History of herpetic keratitis.
* Eye injury within 12 weeks immediately prior to enrollment in this trial.
* Currently enrolled in any clinical trial or participation in any clinical trial within the previous 30 days.
* Other protocol-defined exclusion criteria may apply.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2011-09; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Holden Thomas, OD, Study Director — Alcon Research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 10 investigational centers located in the United States.
Pre-assignment Details: Of the 150 participants enrolled, 3 were exited from the study as screen failures prior to study product dispense. This reporting group includes all randomized and dispensed participants (147).
Period: Overall Study
Arm/Group | AIR OPTIX® COLORS | AIR OPTIX® AQUA
Started | 97 | 50
Completed | 90 | 49
Not Completed | 7 | 1
Not completed — Discomfort | 2 | 0
Not completed — Biomicroscopy | 1 | 0
Not completed — Symptoms and Problems | 1 | 0
Not completed — Unacceptable Subjective Vision | 1 | 0
Not completed — Other Product Related | 1 | 0
Not completed — Unrelated Medical Problem | 0 | 1
Not completed — Other Non-Product Related | 1 | 0

BASELINE CHARACTERISTICS:
Population: The analysis population includes all enrolled participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | AIR OPTIX® COLORS | AIR OPTIX® AQUA | Total
Number analyzed (Participants) | 100 | 50 | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.0 (10.28) | 31.0 (9.91) | 31.0 (10.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 34 | 110
  Male | 24 | 16 | 40

OUTCOME MEASURES:

1. Primary Outcome: Contact Lens-Corrected Distance Monocular Snellen Visual Acuity (VA) (20/30 or Better)
Description: Visual acuity, as assessed for each eye individually. Participant read a distance Snellen chart while wearing study lenses. The percentage of eyes with VA recorded as 20/30 or better is reported. Both eyes contributed to the percentage.
Time Frame: Up to Month 3
Population: The analysis population includes all enrolled and dispensed participants who completed the study. No imputation was used for missing values. Here, "n" is the number of eyes with non-missing values at the specific time point for each arm group, used as the denominator for percentage calculation.
Measure: Number; unit: Percentage of eyes
Units Other Than Participants: Eyes
Arm/Group | AIR OPTIX® COLORS | AIR OPTIX® AQUA
Number analyzed (Participants) | 90 | 49
Number analyzed (Eyes) | 180 | 98
Percentage of eyes
  Dispense (n=180,98) | 100.0 | 100.0
  Week 1 (n=180,98) | 100.0 | 98.0
  Week 2 (n=180,96) | 100.0 | 97.9
  Month 1 (n=180,98) | 100.0 | 100.0
  Month 2 (n=179,98) | 100.0 | 100.0
  Month 3 (n=178,98) | 100.0 | 100.0

2. Secondary Outcome: Subjective Rating of Overall Vision
Description: Overall vision, as rated by the participant on a 10-point scale, with 1 being poor and 10 being excellent. The participant rated both eyes together by providing one single rating.
Time Frame: Up to Month 3
Population: The analysis population includes all enrolled and dispensed participants who completed the study. No imputation was used for missing values. Here, "n" is the number of participants with non-missing values at the specific time point for each arm group.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | AIR OPTIX® COLORS | AIR OPTIX® AQUA
Number analyzed (Participants) | 90 | 49
Units on a scale
  Dispense (n=90,49) | 8.3 (1.7) | 9.5 (0.9)
  Week 1 (n=90,49) | 8.0 (2.1) | 9.4 (0.9)
  Week 2 (n=90,48) | 8.1 (2.0) | 9.4 (0.9)
  Month 1 (n=90,49) | 8.4 (1.9) | 9.3 (0.9)
  Month 2 (n=90,49) | 8.5 (1.8) | 9.3 (1.0)
  Month 3 (n=90,49) | 8.4 (1.8) | 9.3 (1.0)

3. Secondary Outcome: Subjective Rating of Overall Comfort
Description: Overall comfort, as rated by the participant on a 10-point scale, with 1 being poor and 10 being excellent. The participant rated both eyes together by providing one single rating.
Time Frame: Up to Month 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | AIR OPTIX® COLORS | AIR OPTIX® AQUA
Number analyzed (Participants) | 90 | 49
Units on a scale
  Dispense (n=90,49) | 9.1 (1.5) | 9.2 (0.9)
  Week 1 (n=90,49) | 8.3 (1.9) | 9.0 (1.2)
  Week 2 (n=90,48) | 8.6 (1.7) | 9.3 (0.8)
  Month 1 (n=90,49) | 8.4 (1.8) | 8.9 (1.1)
  Month 2 (n=90,49) | 8.5 (1.8) | 8.8 (1.1)
  Month 3 (n=90,49) | 8.6 (1.7) | 8.9 (1.1)

4. Secondary Outcome: Subjective Rating of Overall Handling
Description: Overall handling, as rated by the participant on a 10-point scale, with 1 being difficult and 10 being easy. The participant rated both eyes together by providing one single rating.
Time Frame: Up to Month 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | AIR OPTIX® COLORS | AIR OPTIX® AQUA
Number analyzed (Participants) | 90 | 49
Units on a scale
  Dispense (n=90,49) | 9.3 (1.3) | 9.5 (0.8)
  Week 1 (n=90,49) | 9.4 (1.0) | 9.2 (1.2)
  Week 2 (n=90,48) | 9.4 (1.0) | 9.4 (0.9)
  Month 1 (n=90,49) | 9.5 (0.9) | 9.4 (0.8)
  Month 2 (n=90,49) | 9.4 (1.2) | 9.4 (0.9)
  Month 3 (n=90,49) | 9.4 (1.0) | 9.3 (0.9)

5. Secondary Outcome: Lens Fit (Optimal, Acceptably Loose, Acceptably Tight)
Description: Lens fit, as assessed by the investigator for each eye individually. Lens fit was rated on a 5-point scale: 2=unacceptably loose, 1=acceptably loose, 0=optimal, -1=acceptably tight, -2=unacceptably tight. The combined percentage of lenses assessed as "optimal," "acceptably loose," or "acceptably tight" is reported. Lenses from both eyes contributed to the percentage.
Time Frame: Up to Month 3
Population: as for outcome 1
Measure: Number; unit: Percentage of lenses
Units Other Than Participants: Eyes
Arm/Group | AIR OPTIX® COLORS | AIR OPTIX® AQUA
Number analyzed (Participants) | 90 | 49
Number analyzed (Eyes) | 180 | 98
Percentage of lenses
  Dispense (n=180,98) | 100.0 | 100.0
  Week 1 (n=180,98) | 100.0 | 100.0
  Week 2 (n=180,96) | 100.0 | 100.0
  Month 1 (n=180,98) | 100.0 | 100.0
  Month 2 (n=179,98) | 100.0 | 100.0
  Month 3 (n=180,98) | 100.0 | 100.0

6. Secondary Outcome: Lens Centration (Centered, Slight Decentration)
Description: Lens centration, as assessed by the investigator for each eye individually. Lens centration was rated on a 5-point scale: 0=centered, 1=slight decentration, 2=mild decentration, 3=moderate decentration, 4=severe decentration. The combined percentage of lenses assessed as "centered" or "slight decentration" is reported. Lenses from both eyes contributed to the percentage.
Time Frame: Up to Month 3
Population: as for outcome 1
Measure: Number; unit: Percentage of lenses
Units Other Than Participants: Eyes
Arm/Group | AIR OPTIX® COLORS | AIR OPTIX® AQUA
Number analyzed (Participants) | 90 | 49
Number analyzed (Eyes) | 180 | 98
Percentage of lenses
  Dispense (n=180,98) | 100.0 | 100.0
  Week 1 (n=180,98) | 100.0 | 100.0
  Week 2 (n=180,96) | 100.0 | 100.0
  Month 1 (n=180,98) | 100.0 | 100.0
  Month 2 (n=179,98) | 98.3 | 100.0
  Month 3 (n=180,98) | 100.0 | 100.0

7. Secondary Outcome: Dry Areas/Non-Wetting (None, Very Slight)
Description: Dry areas/non-wetting (i.e., assessment of the disruption of the front surface wettability of the contact lens), as assessed by the investigator for each eye individually. Dry areas/non-wetting was rated on a 5-point scale: 0=none, 1=very slight, 2=slight, 3=moderate, 4=severe. The combined percentage of lenses assessed as "none" or "very slight" is reported. Lenses from both eyes contributed to the percentage.
Time Frame: Up to Month 3
Population: as for outcome 1
Measure: Number; unit: Percentage of lenses
Units Other Than Participants: Eyes
Arm/Group | AIR OPTIX® COLORS | AIR OPTIX® AQUA
Number analyzed (Participants) | 90 | 49
Number analyzed (Eyes) | 180 | 98
Percentage of lenses
  Dispense (n=180,98) | 100.0 | 100.0
  Week 1 (n=180,98) | 100.0 | 99.0
  Week 2 (n=180,96) | 99.4 | 99.0
  Month 1 (n=180,98) | 100.0 | 100.0
  Month 2 (n=179,98) | 100.0 | 100.0
  Month 3 (n=180,98) | 100.0 | 100.0

8. Secondary Outcome: Front Surface Deposits (None, Very Slight)
Description: Front surface deposits on the contact lens, as assessed by the investigator for each eye individually. Front surface deposits were rated on a 5-point scale: 0=none, 1=very slight, 2=slight, 3=moderate, 4=severe. The combined percentage of lenses assessed as "none" or "very slight" is reported. Lenses from both eyes contributed to the percentage.
Time Frame: Up to Month 3
Population: as for outcome 1
Measure: Number; unit: Percentage of lenses
Units Other Than Participants: Eyes
Arm/Group | AIR OPTIX® COLORS | AIR OPTIX® AQUA
Number analyzed (Participants) | 90 | 49
Number analyzed (Eyes) | 180 | 98
Percentage of lenses
  Dispense (n=180,98) | 100.0 | 100.0
  Week 1 (n=180,98) | 96.7 | 98.0
  Week 2 (n=180,96) | 97.8 | 99.0
  Month 1 (n=180,98) | 96.7 | 95.9
  Month 2 (n=179,98) | 97.2 | 98.0
  Month 3 (n=180,98) | 94.4 | 98.0

9. Secondary Outcome: Back Surface Deposits (None, Very Slight)
Description: Back surface deposits on the contact lens, as assessed by the investigator for each eye individually. Back surface deposits were rated on a 5-point scale: 0=none, 1=very slight, 2=slight, 3=moderate, 4=severe. The combined percentage of lenses assessed as "none" or "very slight" is reported. Lenses from both eyes contributed to the percentage.
Time Frame: Up to Month 3
Population: as for outcome 1
Measure: Number; unit: Percentage of lenses
Units Other Than Participants: Eyes
Arm/Group | AIR OPTIX® COLORS | AIR OPTIX® AQUA
Number analyzed (Participants) | 90 | 49
Number analyzed (Eyes) | 180 | 98
Percentage of lenses
  Dispense (n=180,98) | 100.0 | 99.0
  Week 1 (n=180,98) | 100.0 | 100.0
  Week 2 (n=180,96) | 99.4 | 100.0
  Month 1 (n=180,98) | 100.0 | 95.9
  Month 2 (n=179,98) | 99.4 | 100.0
  Month 3 (n=180,98) | 99.4 | 100.0

ADVERSE EVENTS:
Time Frame: Adverse events (AE)s were collected for the duration of the study (4 months). An AE was defined as any untoward medical occurrence in a subject exposed to a test article regardless of causal relationship with the test article.
Description: The analysis population includes all enrolled participants who received study lenses. Adverse events were obtained as solicited comments from the participants and as observations by the Study Investigator as outlined in the study protocol following dispensation of study lenses.
Arm/Group | AIR OPTIX® COLORS | AIR OPTIX® AQUA
Serious Adverse Events (participants affected / at risk) | 0/97 | 0/50
Other Adverse Events (participants affected / at risk) | 0/97 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.